CLINICAL TRIAL: NCT01217632
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled Study of FG-3019 in Subjects With Liver Fibrosis Due to Chronic Hepatitis B Infection
Brief Title: A Study of FG-3019 in Subjects With Liver Fibrosis Due to Chronic Hepatitis B Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to an unexpected prominent effect of entecavir alone in this patient population.
Sponsor: Kyntra Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FGCL-3019-801
Record Dates: First submitted 2010-09-30; First posted 2010-10-08 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Liver Fibrosis Due to Chronic Hepatitis B Infection
Keywords: Connective tissue growth factor (CTGF); human IgG1 monoclonal antibody
MeSH Terms: interventions — pamrevlumab; entecavir; Drugs, Generic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FG-3019 Placebo (Placebo Comparator): Placebo will be administered at 15-45 mg/kg every 3 weeks by IV infusion in a total volume of at least 250 mL in normal saline.
  Interventions: Drug: Placebo; Drug: Entecavir
- FG-3019 (Experimental): FG-3019 at a dose of 15-45 mg/kg will be administered every 3 weeks by IV infusion in a total volume of at least 250 mL in normal saline.
  Interventions: Drug: FG-3019; Drug: Entecavir

INTERVENTIONS:
Drug: FG-3019 — FG-3019 at a dose of 15-45 mg/kg will be administered every 3 weeks by IV infusion in a total volume of at least 250 mL in normal saline.
  Arms: FG-3019
Drug: Placebo — Placebo will be administered every 3 weeks by intravenous (IV) infusion in a total volume of at least 250 mL in normal saline.
  Arms: FG-3019 Placebo
Drug: Entecavir
  Other Names: Entecavir Dispersible (generic)

SUMMARY:
The overall goal of this trial is to evaluate the efficacy of FG-3019 for reversing liver fibrosis in subjects with chronic hepatitis B infection who are beginning antiviral therapy with entecavir. This Phase 2 randomized, double-blind, placebo controlled study will enroll subjects with chronic active hepatitis B infection and liver fibrosis (Ishak score ≥2) who are eligible for antiviral therapy.

ELIGIBILITY:
Inclusion Criteria

* Signed informed consent
* Age of 18 to 75 years, inclusive
* HBsAg positive for ≥24 weeks prior to screening
* Liver fibrosis, confirmed by biopsy and histology
* Willing to use contraception

Exclusion Criteria:

* Female subjects who are pregnant or nursing
* Prior antiviral therapy, with the exception of interferon therapy >6 months prior to Day 1
* Severe heart failure
* Present hepatocellular carcinoma and history of other cancers
* Severe anemia
* Advanced kidney disease
* Immunosuppressive therapy within 24 weeks prior to screening
* Alcohol or drug abuse within the 12 months prior to screening
* Trauma or surgical procedures requiring hospitalization within 8 weeks prior to Day 1
* Planned elective surgery during the study including 9 weeks following the final dose of study drug
* History of allergy against nucleoside analogs or human, humanized, chimeric, or murine monoclonal antibodies
* Inability to cooperate with study personnel or a history of noncompliance to the medical regimen (i.e., subjects who would be expected to comply poorly with the treatment)
* Clinically significant medical or psychiatric condition considered a high risk for participation in an investigational study
* Morbid obesity (body mass index [BMI] >40)
* Inadequate IV access

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2010-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of FG-3019 administered every 3 weeks for 45 weeks on liver fibrosis in subjects with chronic active hepatitis B infection on entecavir therapy | every 3 weeks for 45 weeks

SECONDARY OUTCOMES:
To evaluate the safety, tolerability pharmacokinetic profiles of FG-3019 in the target population | every 3 weeks for 45 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Frank Valone, MD, Study Chair — Kyntra Bio; Mairead Carney, Study Director — Kyntra Bio
Locations (9):
- Hong Kong (6):
  - Queen Mary Hospital, Pokfulam, Hong Kong Island
  - Ruttonjee Hospital, Wan Chai, Hong Kong Island
  - Princess Margaret Hospital, Kowloon, Kowloon
  - Prince of Wales Hospital, Shatin, Kowloon
  - Tuen Mun Hospital, New Territories, New Territories
  - Alice Ho Miu Ling Nethersole Hospital, Tai Po
- Thailand (3):
  - Siriraj Hospital, Siriaj, Bangkok Noi
  - Songklanagarind Hospital, Amphur Hatyai, Changwat Songkhla
  - Maharaj Nakorn Chiang Mai Hospital, Amphur Muang, Chiang Mai